CLINICAL TRIAL: NCT01640015
Title: The Effect of Number of Eating Episodes Per Day on Blood Pressure. A Randomised Controlled Trial
Brief Title: The Effect of Eating Frequency on Blood Pressure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not get ethical approval, therefore study was not initiated
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRO197
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Blood Pressure
Keywords: Blood pressure; eating episode; eating frequency; insulin sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low frequency diet (Experimental): Participants will be assigned to a low frequency diet (fixed energy intake)
  Interventions: Other: dietary intervention
- High frequency diet (Experimental)
  Interventions: Other: dietary intervention

INTERVENTIONS:
Other: dietary intervention — a low frequency diet (3 meals/day) a high frequency diet (9 meals/day)

SUMMARY:
The primary purpose of this study is to identify the effect of meal frequency on blood pressure (BP) levels of individuals.

DETAILED DESCRIPTION:
Migration studies, observational epidemiology and clinical trial data indicate that causes of adverse BP levels are mainly environmental , including lifestyle under which dietary factors play a role. Therefore, lifestyle modification is part of the current American Heart Association recommendations for prevention and control of adverse BP levels.

Although the effects of nutrients and foods on BP have been studied extensively, other dietetic factors such as eating frequency and number of meals in a day have been less thoroughly investigated and warrant further research to explore their possible positive effect on BP.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals aged 35-70 years with prehypertension (systolic/diastolic BP 120-139/80-89 mm Hg) BMI 20-30 kg/m2 non-smoking non alcoholic drinkers

Exclusion Criteria:

* Weight change of ≥ 3kg in the preceding 2 months
* Current smokers
* Substance abuse
* Alcohol intake
* Pregnancy
* Diabetes
* Cardiovascular disease
* Cancer
* Gastrointestinal disease e.g. inflammatory bowel disease or irritable bowel syndrome
* Kidney disease
* Liver disease
* Pancreatitis
* Use of medications including: anti inflammatory drugs or steroids, antihypertensive drugs, cholesterol lowering medication, androgens, phenytoin, erythromycin or thyroid hormones.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01 (Estimated); Primary Completion 2012-01 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 2 weeks for 24 hours through blood pressure monitor
  Participants will be asked to wear BP monitor continuously for one week then return it back either by post or bring it themselves to the center.

SECONDARY OUTCOMES:
Insulin | measured twice during each phase (2 phases)
  biomarkers like: Insulin - Glucose- lipid profile- Free fatty acids- C peptides- HS CRP will be measured regularly during study

CONTACTS AND LOCATIONS:
Locations (1):
- Sir John Michael Center - Hammersmith Hospital, London, United Kingdom